CLINICAL TRIAL: NCT06393296
Title: Melatonin and Secretory Immunoglobulin A (sIgA) Concentration During Lactation, Maternal Determinants and Repercussions
Brief Title: A Study of Melatonin Concentration During Lactation
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Universidade Federal de Goias (Other); University of Wisconsin, Eau Claire (Unknown)
Responsible Party: Principal Investigator, Ganesh Namachivayam, Principal Investigator, Mayo Clinic
Other Study IDs: 23-006493
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Breast milk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breasting Feeding Mothers: New mothers in the immediate postpartum period and breastfeeding their newborn will be asked to collect a sample of breast milk at 14 days postpartum between 6 am and 9 am. In addition to providing a breast milk sample, they will complete a series of questionnaires related to their emotional well-being and lifestyles.

SUMMARY:
This research is being done to understand better how a mother's emotional well-being and lifestyle, such as her levels of stress, fatigue, depression, anxiety, sleep quality, and eating habits, might affect the levels of melatonin and sIgA in her breast milk.

DETAILED DESCRIPTION:
This study aims to learn more about promoting mothers' and babies' health by studying various maternal factors. Gaining a better understanding of the connections between a mother's emotional and physical state and the quality of her breast milk could lead to new recommendations and support strategies to improve the mother's well-being.

Participants will be involved in the study during the immediate postpartum period. They will be asked to provide a 5mL sample of breast milk on day 14 postpartum between 6am and 9am. Participants will be asked to use an orange ambient light during nighttime infant care from the time they come home from the hospital up until the time of breastmilk collection to avoid harsh lighting while providing care for their baby, which may affect melatonin levels.

In addition to breast milk collection, participants will complete a series of questionnaires related to their emotion well-being and lifestyle. These questionnaires will help the research team understand how factors like stress, fatigue, depression, anxiety, sleep, and dietary patterns may be associated with melatonin and sIgA levels in breast milk. Information regarding medications and gestational age of the newborn will be collected from medical records to further assist in data analysis.

ELIGIBILITY:
Inclusion criteria:

* Possess a refrigerator with a freezer or a standalone freezer for sample storage at home.
* Ability to be contacted by telephone.
* Having internet access at home.
* Being in the immediate (0-14 days) postpartum period.
* Currently breastfeeding or planning to breastfeed, regardless of the type.

Exclusion criteria:

* Newborns with congenital malformations.
* Newborns with birth weights less than 2,500g or greater than 4,000g.
* Gestational age less than 37 completed weeks or greater than 42 completed weeks.
* Mothers hospitalized in an intensive care unit (ICU).
* Newborns hospitalized in the neonatal intensive care unit (NICU) or special care nursery (SCN).
* Mothers using sleep aids (e.g., Benadryl, Unisom, Melatonin, Valerian).
* Mothers currently being treated for pharmacologically treated mood and sleep disorders.
* Mothers with acute infections longer than 7 days postpartum. Mothers will be withdrawn from study if antibiotics are taken between 7 and 14 days postpartum.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New mothers receiving care at Mayo Clinic Health System in Eau Claire, Wisconsin.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-10-24 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Melatonin concentration in breast milk | 14 days postpartum
  Melatonin concentration in breast milk samples, reported in picograms per milliliter (pg/mL)
sIgA concentration in breast milk | 14 days postpartum
  concentration in breast milk samples, reported in picograms per milliliter (pg/mL)

SECONDARY OUTCOMES:
Anxiety Symptoms | 14 days postpartum
  Measured using the 14-item Depression, Anxiety and Stress Scale that assesses negative emotional states. Possible total scores range from 0 to 42, with higher scores indicating more negative emotional state and worse outcome.
Depression Symptoms | 14 days postpartum
  Measured using the 10-item Edinburgh Depression Scale (EDS) that assesses depressive symptoms. Possible total scores range from 0 to 30, with higher scores indicating more depressive symptoms and a worse outcome.
Fatigue | 14 days postpartum
  Measured using the 10-item Fatigue Assessment Scale that assesses symptoms of chronic fatigue. Possible total scores range from 10 to 50. A total FAS score < 22 indicates no fatigue, a score ≥ 22 indicates fatigue.
Sleep Quality | 14 days postpartum
  Measured using the The Pittsburgh Sleep Quality Index that assesses the severity of sleep disturbances. Possible scores range from 0 to 21 with higher scores indicating a worse outcome/more severe symptoms of sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Namachivayam, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Health System - Eau Claire, Eau Claire, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Website — https://www.mayoclinic.org
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials